CLINICAL TRIAL: NCT00989365
Title: Effect of Aerobic Training on Psychosocial Morbidity, Symptoms, Airway Inflammation and Autonomic Modulation in Asthmatic Patients
Brief Title: Effect of Aerobic Training on Asthmatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Laboratório de Investigação Médica (Unknown)
Responsible Party: Celso Ricardo Fernandes de Carvalho, School of Medicine, University of São Paulo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Asthmatraining
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Anxiety; Depression; Airway Inflammation
Keywords: Aerobic Exercise; Exercise
MeSH Terms: conditions — Anxiety Disorders; Depression; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient cousenling (Other): Improve medicine use Self control asthma crisis Ambient hygiene
  Interventions: Other: Aerobic training

INTERVENTIONS:
Other: Aerobic training — Treadmill training
  Other Names: Exercise conditioning

SUMMARY:
The investigators hypothesize that aerobic training can reduce anxiety, depression and airway inflammation and those benefits may be related to changes in autonomic system.

DETAILED DESCRIPTION:
One-hundred patients with moderate or severe persistent asthma, age ranging from 20 to 50 years-old recruited after a medical consultation. Asthma diagnosis based on GINA1 and patients were under medical treatment for at least 6-months and considered clinically stable (no crises and changes in medication for at least 30 days). Patients diagnosed with cardiovascular, pulmonary or musculoskeletal diseases impairing exercise training were excluded.

Experimental Design: Patients were studied between 2 medical consultation to avoid changes in medication during the study and patients were randomized (by drawing lots) into either Control or Training groups. CG was submitted to a 4-hour educational program and a breathing exercise program and TG was submitted to the same CG procedures plus an aerobic training program individually based on VO2max. Before and after the intervention, patients performed pulmonary function test and cardiopulmonary exercise testing and as well as fulfilled questionnaires to quantify asthma specific HRQL and anxiety and depression levels. Asthma daily symptoms were evaluated monthly.

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years old
* moderate and severe asthma

Exclusion Criteria:

* other pulmonary or cardiovascular disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
psychosocial morbidity and airway inflammation | 3 months

SECONDARY OUTCOMES:
autonomic modulation, aerobic capacity, pulmonary function | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, PhD, Study Chair — School of Medicine, University of São Paulo
Locations (1):
- Clinical Hospital, School of Medicine, University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Fanelli A, Cabral AL, Neder JA, Martins MA, Carvalho CR. Exercise training on disease control and quality of life in asthmatic children. Med Sci Sports Exerc. 2007 Sep;39(9):1474-80. doi: 10.1249/mss.0b013e3180d099ad. PMID 17805077
- [Derived] Mendes FA, Goncalves RC, Nunes MP, Saraiva-Romanholo BM, Cukier A, Stelmach R, Jacob-Filho W, Martins MA, Carvalho CR. Effects of aerobic training on psychosocial morbidity and symptoms in patients with asthma: a randomized clinical trial. Chest. 2010 Aug;138(2):331-7. doi: 10.1378/chest.09-2389. Epub 2010 Apr 2. PMID 20363839